CLINICAL TRIAL: NCT02129855
Title: Metabolic Costs of Daily Activities in Older Adults
Acronym: CHORES-XL
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Wake Forest University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201501057-N; 5R01AG042525-05 (NIH); 087-2013 (Other: Univeristy of Florida); OCR15164 (Other: University of Florida)
Record Dates: First submitted 2014-02-28; First posted 2014-05-02 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Functional Limitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The work will evaluate the metabolic costs for daily activities across the lifespan and evaluate the influence of having functional impairments.

DETAILED DESCRIPTION:
The work will evaluate the metabolic costs for daily activities across the lifespan and evaluate the influence of having functional impairments. The project will simultaneously conduct a cross-sectional and a case-control study. The primary aim will investigate cross-sectional association between older age and the energy expenditure of daily activities by recruiting approximately 25 adults in each of 7 age groups (20-30,30-40,40-50,50-60,60-70,70-80,80+) for a total of 180 individuals. A secondary aim will investigate the effect of functional impairments on the energy expenditure of daily activities by conducting a case-control study. An additional 25 older adults with functional impairment will be recruited in each age decade (60-70, 70-80, and 80+ years old) to accomplish this aim. Additional outcomes will evaluate rating of perceived exertion differences in daily activities. A tertiary aim will investigate using accelerometers to predict the metabolic costs of daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Age 20+ years old
* Community dwelling adults without significant health issues
* Willingness to undergo all testing procedures
* Weight stable for at least three months
* Able to understand and speak English

Exclusion Criteria:

* Failure to provide informed consent
* A 10% enrollment limit will be applied to avid exercisers in each age decade. Avid exercises will be defined as doing structured exercise 3 or more days per week (e.g. jogging, sports etc., walkers will be permitted in the study). Based on our experience, avid exercisers volunteer for this type of research at a high rate and thus the investigators will limit these individuals to prevent a biased comparison
* Use of walker (use of a cane is permitted)
* Lower extremity amputation
* Develops chest pain or severe shortness of breath during physical stress
* Post-stroke syndrome causing ambulatory deficits (other stroke survivors permitted)
* Pacemaker
* Needs assistance with basic activities of daily living: feeding, dressing, continence, bathing, toileting, and transferring from a bed to a chair or from a chair to walking
* Lives in a nursing home; persons living in assisted or independent housing are not excluded
* For adults over the age of 60: >2 errors on the Short, portable mental status questionnaire administered after written informed consent
* Excessive alcohol or substance abuse within six months or consumption of >14 alcohol drinks/week
* For women who are child-bearing age (up to 62 years of age): pregnant or breast-feeding
* Participation in a structured weight loss program or fad diet in the last month;
* Weight reduction surgery in the past year
* Known neuromuscular disorder (Rhabdomyolysis, Myasthenia Gravis, Ataxia, Apraxia, post-polio syndrome, mitochondrial myopathy, chronic fatigue syndrome etc.)
* Diagnosed neuropathy that causes pain
* Symptomatic peripheral arterial disease
* Unable to communicate because of severe hearing loss or speech disorder
* Severe visual impairment, which would preclude completion of the assessments
* Progressive, degenerative neurologic disease, e.g., Parkinson's Disease, Multiple Sclerosis, Amyotrophic lateral sclerosis
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, active inflammatory disease; self-reported severe osteoarthritis
* Terminal illness, as determined by the participant
* Severe pulmonary disease, requiring the use of supplemental oxygen or steroid therapy
* Severe cardiac disease, including New York Heart Association Class III or IV congestive heart failure, clinically significant aortic stenosis, recent history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Other significant comorbid disease discovered during medical screening, e.g. renal failure on hemodialysis, psychiatric disorder (e.g. bipolar, schizophrenia); chronic fatigue syndrome etc…
* Liver diseases: chronic hepatitis, an inflammatory disease, or cirrhosis
* Pregnancy. Participants within childbearing age will have a pregnancy test.
* Contraindications to graded exercise testing according to the American Thoracic Society:
* Acute myocardial infarction (<6 months since event)
* Unstable angina
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise
* Syncope
* Active endocarditis
* Acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolus or pulmonary infarction
* Thrombosis of lower extremity
* Suspected dissecting aneurysm
* Uncontrolled asthmas
* Pulmonary edema
* Room air desaturation at rest < 85%
* Respiratory failure
* Acute non cardiopulmonary disorder that may affect exercise performance

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling population
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2014-07; Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
MET value | Participants will attend up to 4 visits within one month of enrollment to attain these data
  MET value of physical activities defined as the oxygen uptake (VO2 = milliliter• min-1•kg-1) during a steady state rate expressed as a function 3.5 milliliter• min-1•kg-1.
Metabolic economy | Participants will attend up to 4 visits within one month of enrollment to attain these data
  Metabolic economy is the energy expended for a given work rate.
Relative metabolic cost to peak energy expenditure | Participants will attend up to 4 visits within one month of enrollment to attain these data
  Relative metabolic cost is function of peak oxygen consumption
Relative metabolic cost to resting energy expenditure | Participants will attend up to 4 visits within one month of enrollment to attain these data
  Relative metabolic cost as a function of resting

SECONDARY OUTCOMES:
Rating of perceived exertion | Participants will attend up to 4 visits within one month of enrollment to attain these data
  Ratings of perceived exertion will be collected during all activities. Investigators will use the Category Ratio scale-10 scale developed by Borg in 1982.

OTHER OUTCOMES:
Accelerometer signals to predict of energy expenditure | Participants will attend up to 4 visits within one month of enrollment to attain these data
  A tertiary outcome is to validate body worn monitors (e.g. accelerometers) to estimate the type and intensity of activity for accurate estimation of energy expenditure. A predicted metabolic equivalent value will be estimated for each activity.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Manini, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Institute on Aging Clinical and Translational Research Building, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: University of Florida Institute on Aging — http://aging.ufl.edu/